CLINICAL TRIAL: NCT03089944
Title: A Single Arm, Open-label Study to Evaluate the Efficacy and Safety of Glecaprevir (GLE)/Pibrentasvir (PIB) in Treatment Naïve Adults With Chronic Hepatitis C Virus (HCV) Genotype 1-6 Infection and Compensated Cirrhosis
Brief Title: A Study of Glecaprevir (GLE)/Pibrentasvir (PIB) in Treatment-Naive Adults With Chronic Hepatitis C Virus (HCV) Genotype 1-6 Infection and Compensated Cirrhosis
Acronym: EXPEDITION-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-135; 2016-004967-38 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2017-03-22; First posted 2017-03-24 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C Virus (HCV); Glecaprevir; Pibrentasvir; Treatment Naïve; Cirrhosis; Compensated Cirrhosis; Genotype (GT) 1-6; Pangenotypic; Chronic Hepatitis C Virus (HCV)
MeSH Terms: conditions — Hepatitis C; Fibrosis; Hepatitis C, Chronic | interventions — glecaprevir and pibrentasvir; glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 weeks (Experimental): Glecaprevir (GLE)/Pibrentasvir (PIB) 300 mg/120 mg once daily (QD) for 8 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Tablet
  Other Names: ABT-493; ABT-530

SUMMARY:
A Phase 3b, single arm, open-label, multicenter study in treatment naïve adults with chronic HCV infection and compensated cirrhosis to assess the safety of 8 weeks of treatment with glecaprevir/pibrentasvir and to demonstrate the efficacy of the sustained virologic response 12 weeks post dosing (SVR12) rates of 8 weeks of treatment with glecaprevir/pibrentasvir compared to the historical SVR12 rates of 12 weeks of treatment with glecaprevir/pibrentasvir.

ELIGIBILITY:
Inclusion Criteria:

* Screening laboratory result indicating Hepatitis C Virus (HCV) Genotype (GT) 1-6 infection.
* Positive plasma HCV antibody and HCV RNA viral load greater than or equal to 1000 IU/mL at Screening.
* Treatment-naive to any approved or investigational anti-HCV medication.
* Participant must be documented as cirrhotic, with a Child-Pugh score of less than or equal to 6.

Exclusion Criteria:

* Female participant who is pregnant, breastfeeding or is considering becoming pregnant during the study, or for approximately 30 days after the last dose of study drug.
* Any current or historical clinical evidence of decompensated cirrhosis.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg), HBV deoxyribonucleic acid > lower limit of quantification (LLOQ) in subjects with isolated positive antibody to hepatitis B core antigen (anti-HBc) (i.e., negative HBsAg and anti-hepatitis B),or anti human immunodeficiency virus antibody (HIV Ab).
* HCV genotype performed by the central laboratory during screening indicating co-infection with more than one HCV genotype.
* History of suspected or confirmed hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (113):
- United States (40):
  - St. Josephs Hosp and Med Ctr /ID# 162762, Phoenix, Arizona
  - Mayo Clinic Arizona /ID# 162314, Phoenix, Arizona
  - Liver Wellness Center /ID# 162244, Little Rock, Arkansas
  - Felizarta /ID# 162295, Bakersfield, California
  - VA Long Beach Healthcare System /ID# 162298, Long Beach, California
  - Usc /Id# 162248, Los Angeles, California
  - Kaiser Permanente - San Diego (Palm Ave) /ID# 162289, San Diego, California
  - Stanford University School of Med /ID# 162209, Stanford, California
  - Cedars-Sinai Medical Center - West Hollywood /ID# 162313, West Hollywood, California
  - University of Miami /ID# 162210, Miami, Florida
  - Triple O Research Institute /ID# 162300, West Palm Beach, Florida
  - Piedmont Hospital /ID# 162646, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 162208, Chicago, Illinois
  - Unity Point Health /ID# 162247, Des Moines, Iowa
  - The University of Iowa Hospita /ID# 162214, Iowa City, Iowa
  - University of Louisville /ID# 162242, Louisville, Kentucky
  - Louisiana Research Ctr. LLC /ID# 162567, Shreveport, Louisiana
  - Mercy Medical Center /ID# 162291, Baltimore, Maryland
  - Mayo Clinic - Rochester /ID# 162251, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 162241, Jackson, Mississippi
  - CHI Health Alegent Creighton /ID# 162286, Omaha, Nebraska
  - Univ Nebraska Med Ctr /ID# 162285, Omaha, Nebraska
  - Rnjms /Id# 162213, Newark, New Jersey
  - Weill Cornell Medical College /ID# 161051, New York, New York
  - Icahn School of Med Mt. Sinai /ID# 162294, New York, New York
  - Montefiore Medical Center /ID# 162312, The Bronx, New York
  - James J. Peters VA Medical Center /ID# 162644, The Bronx, New York
  - Duke University Medical Center /ID# 162299, Durham, North Carolina
  - Cumberland Research Assoc /ID# 162212, Fayetteville, North Carolina
  - Carolinas Center for Liver Dis /ID# 162569, Statesville, North Carolina
  - University Hospitals Cleveland /ID# 162243, Cleveland, Ohio
  - Cleveland Clinic /ID# 162570, Cleveland, Ohio
  - Osuchs /Id# 162284, Tulsa, Oklahoma
  - Lehigh Valley Health Network /ID# 162603, Allentown, Pennsylvania
  - Center for Liver Diseases, Oakland /ID# 162568, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr /ID# 162211, Nashville, Tennessee
  - Texas Digestive Disease Consul /ID# 162648, Dallas, Texas
  - University of Texas Health /ID# 162288, Houston, Texas
  - Virginia Commonwealth Univ /ID# 162215, Richmond, Virginia
  - Univ of Wisconsin Hosp/Clinics /ID# 162645, Madison, Wisconsin
- Bulgaria (4):
  - Tokuda Hospital Sofia /ID# 163422, Sofia
  - DCC Fokus-5 - LZIP /ID# 163338, Sofia
  - Univ Hosp for Active Treat /ID# 163330, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 163332, Sofia
- Canada (5):
  - University of Calgary /ID# 161185, Calgary, Alberta
  - Percuro Clinical Research, Ltd /ID# 161184, Victoria, British Columbia
  - Qe Ii Hsc /Id# 161178, Halifax, Nova Scotia
  - The Ottawa Hospital Research /ID# 161179, Ottawa, Ontario
  - Toronto General Hospital /ID# 161182, Toronto, Ontario
- Czechia (3):
  - Research Site s.r.o /ID# 163020, Pilsen
  - KlinMed s.r.o. /ID# 162893, Prague
  - Institut Klinicke a Experimeth /ID# 162900, Prague
- France (6):
  - CHR Orleans - Hopital de la Source /ID# 163072, Orléans, Centre-Val de Loire
  - Hôpital Purpan /ID# 163065, Toulouse, Haute-Garonne
  - CHU Amiens Picardie /ID# 163071, Amiens, Somme
  - CHU Estaing /ID# 163058, Clermont-Ferrand
  - Hospital Henri Mondor /ID# 163061, Créteil
  - Hopital de la Croix Rousse /ID# 163073, Lyon
- Greece (4):
  - General Hospital of Athens Laiko /ID# 162786, Athens, Attica
  - General and Oncology Hospital /ID# 162784, Kifissia
  - Reg Gen Univ Hosp Larissa /ID# 162783, Larissa
  - Bioclinic Thessaloniki /ID# 162785, Thessaloniki
- Hungary (2):
  - Budai Hepatologiai Centrum /ID# 166511, Budapest
  - Szent Janos Korhaz /ID# 166542, Budapest
- Ireland (3):
  - St. James's Hospital /ID# 162619, Dublin, Dublin
  - Beaumont Hospital /ID# 162618, Dublin
  - St Vincent's Hospital /ID# 162617, Dublin
- Israel (4):
  - Tel Aviv Sourasky Medical Ctr /ID# 162185, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 162023, Haifa
  - The Lady Davis Carmel MC /ID# 162017, Haifa
  - Sheba Medical Center /ID# 162028, Ramat Gan
- Italy (5):
  - Universita della Campania Luigi Vanvitelli /ID# 162337, Napoli, Campania
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 162335, Bologna, Emilia-Romagna
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 162340, Milan, Lombardy
  - Istituto Clinico Humanitas /ID# 162336, Rozzano, Milano
  - Polo Universitario Luigi Sacco /ID# 162339, Milan
- Poland (4):
  - Centrum Badan Klinicznych, Przychodnia Badan Klinicznych /ID# 162760, Wroclaw, Lower Silesian Voivodeship
  - HepID - Diagnostyka I Terapia /ID# 162761, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczn /ID# 162757, Bialystok
  - ID Clinic /ID# 162759, Mysłowice
- Portugal (4):
  - Centro Hosp de Lisboa Central /ID# 163770, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 163785, Lisbon
  - Centro Hospitalar do Porto EPE /ID# 163765, Porto
  - Centro Hospitalar de Sao Joao /ID# 163766, Porto
- Puerto Rico (3):
  - GHGCPR Research Institute /ID# 162608, Ponce
  - Instituto de Investigacion Cientifica del Sur /ID# 162566, Ponce
  - Klinical Investigations Group /ID# 162565, San Juan
- Romania (5):
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals /ID# 163484, Sector 2, București
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals /ID# 164449, Sector 2, București
  - Institutul Clinic Fundeni /ID# 163479, Sector 2, București
  - Institutul Clinic Fundeni /ID# 163500, Sector 2, București
  - Institutul Nat. de Boli Infectioase /ID# 163488, Bucharest
- Russia (5):
  - LLC Medical Company Hepatolog /ID# 161998, Samara, Samara Oblast
  - CBSI Central scientific and research institute of epidemiology /ID# 161996, Moscow
  - Central Clinical Hospital of R /ID# 163434, Moscow
  - Stavropol State Medical Univ /ID# 161999, Stavropol
  - RSAHI Consulting and Diagnostic Centre /ID# 161995, Tyumen
- Spain (5):
  - Hospital Parc de Salut del Mar /ID# 162198, Barcelona
  - Hospital Univ Vall d'Hebron /ID# 162199, Barcelona
  - Hospital Universitario Reina S /ID# 162200, Córdoba
  - Hospital Donostia /ID# 162197, Donostia / San Sebastian
  - Hospital Univ Central Asturias /ID# 162195, Oviedo
- Taiwan (3):
  - China Medical University Hosp /ID# 162950, Taichung, Taichung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 162949, Kaohsiung City
  - Taipei Veterans General Hosp /ID# 162776, Taipei
- United Kingdom (5):
  - Basildon University Hospital /ID# 162616, Basildon, Essex
  - The Royal Free Hospital /ID# 162614, London, London, City of
  - North Manchester General /ID# 163945, Crumpsall
  - Western General Hospital /ID# 162612, Edinburgh
  - Queens Medical Centre /ID# 162615, Nottinghamshire
- Vietnam (3):
  - National Hospital of Tropical Diseases /ID# 167974, Hanoi
  - Hoa Hao Medic Co. Ltd. /ID# 168178, Ho Chi Minh City
  - Tropical Diseases Hospital /ID# 168211, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Brown RS Jr, Buti M, Rodrigues L, Chulanov V, Chuang WL, Aguilar H, Horvath G, Zuckerman E, Carrion BR, Rodriguez-Perez F, Urbanek P, Abergel A, Cohen E, Lovell SS, Schnell G, Lin CW, Zha J, Wang S, Trinh R, Mensa FJ, Burroughs M, Felizarta F. Glecaprevir/pibrentasvir for 8 weeks in treatment-naive patients with chronic HCV genotypes 1-6 and compensated cirrhosis: The EXPEDITION-8 trial. J Hepatol. 2020 Mar;72(3):441-449. doi: 10.1016/j.jhep.2019.10.020. Epub 2019 Nov 2. PMID 31682879

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 343 participants were enrolled and received ≥ 1 dose of study drug.
Groups:
- Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks: GLE/PIB 300 mg/120 mg once daily (QD) for 8 weeks.
Period: Overall Study
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Started | 343
Completed | 331
Not Completed | 12
Not completed — Lost to Follow-up | 8
Not completed — Withdrew Consent | 2
Not completed — Adverse Event | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of study drug were included.
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.61 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 300
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 285
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Hepatitis C Virus (HCV) Genotype (GT) 1,2,4,5 and 6-infected Participants in the Per Protocol (PP) Population
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (<LLOQ; less than 15 IU/mL) 12 weeks after the last dose of study drug. Efficacy of the 8-week treatment duration compared to the historical 12-week treatment duration was demonstrated if the lower bound of the 2-sided 95% confidence interval (CI) for the percentage of participants with HCV GT1, GT2, GT4, GT5, or GT6 infection in the 8 week treatment duration achieving SVR12 was greater than 94% in the PP population. Efficacy analyses were performed following a fixed-sequence testing procedure to control the type I error rate. The percentage of participants achieving SVR12 was summarized with a 2-sided 95% CI, calculated using the normal approximation to the binomial distribution. If the number of participants who failed to achieve SVR12 rate was less than 5, the Wilson's score method was used to calculate the CI.
Time Frame: 12 weeks after last dose of study drug
Population: Per Protocol (PP) Population: All participants who received at least one dose of study drug, with the exception of participants who experienced breakthrough, or prematurely discontinued treatment prior to Week 8, or had no HCV RNA value in the SVR12 visit window or later.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 274
percentage of participants | 100 [98.6 to 100.0]

2. Primary Outcome: Percentage of Participants With SVR12 in HCV GT 1,2,4,5 and 6-infected Participants in the Intent-To-Treat (ITT) Population
Description: SVR12 was defined as HCV RNA level less than the LLOQ (less than 15 IU/mL) 12 weeks after the last dose of study drug. Efficacy of the 8-week treatment duration compared to the historical 12-week treatment duration was demonstrated if the lower bound of the 2-sided 95% CI for the percentage of participants with HCV GT1, GT2, GT4, GT5, or GT6 infection in the 8 week treatment duration achieving SVR12 was greater than 93% in the ITT population. Primary efficacy analyses were performed following a fixed-sequence testing procedure to control the type I error rate. The percentage of participants achieving SVR12 was summarized with a 2-sided 95% CI, calculated using the normal approximation to the binomial distribution. If the number of participants who failed to achieve SVR12 rate was less than 5, the Wilson's score method was used to calculate the CI.
Time Frame: 12 weeks after last dose of study drug
Population: Intent to treat (ITT) population: Participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 280
percentage of participants | 98.2 [96.7 to 99.8]

3. Secondary Outcome: Percentage of Participants With SVR12 in HCV GT1-6-infected Participants in the PP Population
Description: SVR12 was defined as HCV RNA level less than the LLOQ (less than 15 IU/mL) 12 weeks after the last dose of study drug. Efficacy of the 8-week treatment duration compared to the historical 12-week treatment duration was demonstrated if the lower bound of the 2-sided 95% CI for the percentage of participants with HCV GT1, GT2, GT3, GT4, GT5, or GT6 infection in the 8 week treatment duration achieving SVR12 was greater than 94% in the PP population. These efficacy analyses were performed only if success was demonstrated for both primary efficacy analyses, following a fixed-sequence testing procedure.
Time Frame: 12 weeks after last dose of study drug
Population: PP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 335
percentage of participants | 99.7 [98.3 to 99.9]

4. Secondary Outcome: Percentage of Participants With SVR12 in HCV GT1-6-infected Participants in the ITT Population
Description: SVR12 was defined as HCV RNA level less than the LLOQ (less than 15 IU/mL) 12 weeks after the last dose of study drug. Efficacy of the 8-week treatment duration compared to the historical 12-week treatment duration was demonstrated if the lower bound of the 2-sided 95% CI for the percentage of participants with HCV GT1, GT2, GT3, GT4, GT5, or GT6 infection in the 8 week treatment duration achieving SVR12 was greater than 93% in the ITT population. These efficacy analyses were performed only if success was demonstrated for both primary efficacy analyses, following a fixed-sequence testing procedure.
Time Frame: 12 weeks after the last dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 343
percentage of participants | 97.7 [96.1 to 99.3]

5. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure in the ITT Population
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: 8 weeks on treatment
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 343
percentage of participants | 0 [0.0 to 1.1]

6. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment as planned (defined as study drug duration ≥ 52 days for participants assigned to 8 weeks of treatment) and with HCV RNA levels < LLOQ at the end of treatment excluding participants who had been reinfected.
Time Frame: Up to 12 weeks after the last dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 336
percentage of participants | 0.3 [0.1 to 1.7]

7. Secondary Outcome: Percentage of HCV GT3-infected Participants Who Achieved SVR12 in the PP Population
Description: SVR12 was defined as HCV RNA level less than the LLOQ (less than 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of study drug
Population: PP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 61
percentage of participants | 98.4 [91.3 to 99.7]

8. Secondary Outcome: Percentage of HCV GT3-infected Participants Who Achieved SVR12 in the ITT Population
Description: SVR12 was defined as HCV RNA level less than the LLOQ (less than 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks
Number analyzed (Participants) | 63
percentage of participants | 95.2 [86.9 to 98.4]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were defined as any adverse event with an onset date that was on or after the first dose of study drug and no more than 30 days after the last dose of study drug.
Groups:
- Glecaprevir (GLE)/Pibrentasvir (PIB): GLE/PIB 300 mg/120 mg once daily (QD) for 8 weeks.
Arm/Group | Glecaprevir (GLE)/Pibrentasvir (PIB)
All-Cause Mortality (participants affected / at risk) | 0/343
Serious Adverse Events (participants affected / at risk) | 6/343
Other Adverse Events (participants affected / at risk) | 82/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir (GLE)/Pibrentasvir (PIB) (N=343)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir (GLE)/Pibrentasvir (PIB) (N=343)
NAUSEA (Gastrointestinal disorders) | 19 (19)
FATIGUE (General disorders) | 30 (30)
HEADACHE (Nervous system disorders) | 28 (28)
PRURITUS (Skin and subcutaneous tissue disorders) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03089944/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03089944/SAP_001.pdf